CLINICAL TRIAL: NCT06993441
Title: Effects of Music on Pain, Anxiety and Stress Levels in Cancer Patients Receiving Radiotherapy
Brief Title: Music and Symptom Relief in Radiotherapy Patient
Acronym: MUSİC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Duygu Akbas Uysal, Dr., Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1150
Record Dates: First submitted 2025-05-13; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Music Therapy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Participants in this group will listen to MusICure music through speakers for 30 minutes during each radiotherapy session. The intervention is designed to provide a calming auditory experience to reduce anxiety and improve comfort during treatment.
  Interventions: Behavioral: Experimantal group
- control group (Experimental)
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: Experimantal group — Participants in the experimental group listened to MusICure music via speakers for 30 minutes during each radiotherapy session. The intervention was administered concurrently with radiotherapy and aimed to reduce anxiety and emotional distress.
  Arms: Experimental Arm
Behavioral: control group — No intervention
  Arms: control group

SUMMARY:
This randomized controlled study aims to evaluate the effects of music therapy administered during radiotherapy sessions on pain, stress, and anxiety levels in cancer patients. The intervention involves playing Musicure, a therapeutic music track, for 30 minutes via speakers during radiotherapy. The study includes two groups: an intervention group receiving music therapy and a control group receiving standard care without music.

Participants' pain levels were assessed using the Visual Analog Scale (VAS), while anxiety and stress levels were measured using the Face Anxıety Subscale ( FAS).

A total of 120 adult cancer patients undergoing outpatient radiotherapy at Tınaztepe Unıversty were included. The study was conducted under the supervision of Dr. Öğr. Üyesi [Duygu AKBAŞ UYSAL (Principal Investigator) and co-researchers Prof.Dr Fsun ŞENUZUN AYKAR, Prof.Dr Zümra ARICAK ALICIKUŞ The research complies with ethical standards and has received approval from [insert name of ethics committee].

This study investigates a low-cost, non-pharmacological intervention that has the potential to improve symptom management and quality of life in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study,
* 18 years of age and older,
* No hearing problems,
* No communication and speech problems

Exclusion Criteria:

* Those diagnosed with psychiatric and neurological diseases,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Pain Level | Baseline (before radiotherapy on Day 1) and immediately after the radiotherapy session on Day 1.
  Changes in pain levels were assessed using the Visual Analog Scale (VAS) immediately before and after a single radiotherapy session. The VAS score ranges from 0 (no pain) to 10 (worst possible pain).

SECONDARY OUTCOMES:
anxiety level | Baseline (before radiotherapy on Day 1) and immediately after the radiotherapy session on Day 1.
  Changes in anxiety levels were assessed using the Facial Anxiety Scale (FAS), a visual scale ranging from 0 (no anxiety) to 5 (severe anxiety), immediately before and after a single radiotherapy session.

CONTACTS AND LOCATIONS:
Locations (1):
- Tinazetepe Bayrakli Hospital, Izmir, İzmir, Turkey (Türkiye)